CLINICAL TRIAL: NCT05685966
Title: Retrospective Study of COVID-19 on Reproductive Function and Assisted Reproductive Technology Pregnancy Outcome in China
Brief Title: Retrospective Study of COVID-19 on Reproductive Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Bing Yao, Professor, Jinling Hospital, China
Other Study IDs: Retrospective study of COVID19
Record Dates: First submitted 2023-01-13; First posted 2023-01-17 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19; Reproductive function; Sustained pregnancy rate
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum, seminal plasma, sperm, follicular Fluid, granule cells, embryo culture medium, endometrial tissue, villi and decidual tissue if abortion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile couples from the research center who visited for fertility disorders: Infertile couples infected or not infected with COVID-19 were included.This is an observational study with no interventions.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This multi-center, retrospective cohort study aimed to determine which factors are associated with ongoing pregnancy rates in infertile patients received ART treatments during the current outbreak of COVID-19 infection.Couples who underwent IVF-ET/ICSI-ET/FET due to infertility in the department of Reproductive Medicine from 2022-11-23 to 2023-01-07 were included. Patients who were infected with Coronavirus were observation groups; the infection status and clinical outcome were tracked. Patients who were not infected with Coronavirus were control groups.

DETAILED DESCRIPTION:
In this multi-center, retrospective cohort study, we included patients who underwent IVF-ET/ICSI-ET/FET due to infertility in the department of Reproductive Medicine from 2022-11-23 to 2023-01-07. Patients who were infected with Coronavirus were observation groups; the infection status and clinical outcome were tracked. Patients who were not infected with Coronavirus were control groups. We compared different parameters between two groups. The primary outcome was ongoing pregnancy rate. Basic information about patients' menstruation, sexual desire, and sexual function were collected from Medical record system. Other information about patients' vaccination status, symptoms related to viral infection were collected by telephone follow ups. Susceptibility indicators to COVID-19 infection including fasting blood glucose, insulin, blood lipids, alpha-function, renin-angiotensinase, I-aldosterone were obtained . Reproductive function indices AMH, INHB, sex hormones, follicle retrieval rate, Gn days, total Gn, endometrial thickness, the incidence of OHSS, semen quality, oocyte maturation rate, fertilization rate, qualified embryo rate, blastocyst formation rate, and other laboratory indices of both men and women were also collected . Assisted pregnancy outcome: clinical pregnancy rate, embryo implantation rate, early abortion rate, ongoing pregnancy rate, and other clinical indicators were analyzed to determine whether there is deference in clinical outcomes between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with infertility
* Patients with IVF-ET/ICSI-ET/FET from 2022/11/23 to 2023/01/07

Exclusion Criteria:

* Patients with contraindications to pregnancy or assisted reproductive technology

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Failure to establish a clinical pregnancy after 12 months of regular unprotected intercourse, or due to impaired fertility of the individual or his or her partner, is termed infertility.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 3 months
  If the fetal sac, fetal bud, and primitive fetal heartbeat are found by vaginal B-ultrasound examination 55-65 days after embryo transfer, the diagnosis of ongoing pregnancy will be made.

SECONDARY OUTCOMES:
Clinical and laboratory indicators related to male and female reproductive function | 3 months
  AMH, INB, sex hormone, follicle output rate, Gn days, total Gn, endometrial thickness on the embryo transfer day, semen quality; Oocyte maturation rate, fertilization rate, high-level embryo rate, blastocyst formation rate
Outcome indicators of assisted pregnancy | 3 months
  Embryo implantation rate, early abortion rate, ongoing pregnancy rate, incidence of OHSS

OTHER OUTCOMES:
Coagulation index | 3 months
  D-dimer
Indicators of susceptibility to COVID-19 infection | 3 months
  blood lipid, blood sugar, insulinand thyroid function
Oxidative stress index | 3 months
  fingertip pulse oxygen saturation
SAS Anxiety Scale | 3 months
  SAS Anxiety Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bing Yao, PHD, Study Chair — Department of Reproductive Medicine, Jinling Hospital; Li Chen, PHD, Study Director — Department of Reproductive Medicine, Jinling Hospital; Xiaojie Huang, PHD, Principal Investigator — Department of Reproductive Medicine, Xuzhou Maternal and Child Health Care Hospital; Jiayi Ding, PHD, Principal Investigator — Department of Reproductive Medicine, Nantong Maternal and Child Health Care Hospital; Qin Sun, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Meiling Li, PHD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Cheng Zhou, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Xi Chen, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Yuming Feng, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Juanjuan Xu, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Haiyan Fu, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Cencen Wang, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Hong Zhang, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Lu Zheng, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Yuxiu Liu, PHD, Principal Investigator — Department of Critical Care Medicine, Jinling Hospital; Xiaofang Tan, MD, Principal Investigator — Department of Reproductive Medicine, Nantong Maternal and Child Health Care Hospital; Yunxia Zhu, MD, Principal Investigator — Department of Reproductive Medicine, Xuzhou Maternal and Child Health Care Hospital; Jueraitetibaike Kadiliya, PHD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Zhichan Zou, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital
Locations (3):
- China (3):
  - Department for Reproductive Medicine, Jinling Hospital, Nanjing, Jiangsu
  - Department of Reproductive Medicine, Nantong Maternal and Child Health Care Hospital, Nantong, Jiangsu
  - Department of Reproductive Medicine, Xuzhou Maternal and Child Health Care Hospital, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Chu H, Zhou J, Wong BH, Li C, Chan JF, Cheng ZS, Yang D, Wang D, Lee AC, Li C, Yeung ML, Cai JP, Chan IH, Ho WK, To KK, Zheng BJ, Yao Y, Qin C, Yuen KY. Middle East Respiratory Syndrome Coronavirus Efficiently Infects Human Primary T Lymphocytes and Activates the Extrinsic and Intrinsic Apoptosis Pathways. J Infect Dis. 2016 Mar 15;213(6):904-14. doi: 10.1093/infdis/jiv380. Epub 2015 Jul 22. PMID 26203058
- [Background] Xia W, Shao J, Guo Y, Peng X, Li Z, Hu D. Clinical and CT features in pediatric patients with COVID-19 infection: Different points from adults. Pediatr Pulmonol. 2020 May;55(5):1169-1174. doi: 10.1002/ppul.24718. Epub 2020 Mar 5. PMID 32134205
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Bobrova L, Kozlovskaya N, Korotchaeva Y, Bobkova I, Kamyshova E, Moiseev S. Microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome (MicroCLOTS): a new variant of thrombotic microangiopathy? Crit Care Resusc. 2020 Sep;22(3):284. doi: 10.1016/S1441-2772(23)00399-X. No abstract available. PMID 32900338
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Danzi GB, Loffi M, Galeazzi G, Gherbesi E. Acute pulmonary embolism and COVID-19 pneumonia: a random association? Eur Heart J. 2020 May 14;41(19):1858. doi: 10.1093/eurheartj/ehaa254. No abstract available. PMID 32227120
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Wu M, Ma L, Xue L, Zhu Q, Zhou S, Dai J, Yan W, Zhang J, Wang S. Co-expression of the SARS-CoV-2 entry molecules ACE2 and TMPRSS2 in human ovaries: Identification of cell types and trends with age. Genomics. 2021 Nov;113(6):3449-3460. doi: 10.1016/j.ygeno.2021.08.012. Epub 2021 Aug 18. PMID 34418496
- [Background] Boudry L, Essahib W, Mateizel I, Van de Velde H, De Geyter D, Pierard D, Waelput W, Uvin V, Tournaye H, De Vos M, De Brucker M. Undetectable viral RNA in follicular fluid, cumulus cells, and endometrial tissue samples in SARS-CoV-2-positive women. Fertil Steril. 2022 Apr;117(4):771-780. doi: 10.1016/j.fertnstert.2021.12.032. Epub 2022 Jan 1. PMID 35272846
- [Background] Li K, Chen G, Hou H, Liao Q, Chen J, Bai H, Lee S, Wang C, Li H, Cheng L, Ai J. Analysis of sex hormones and menstruation in COVID-19 women of child-bearing age. Reprod Biomed Online. 2021 Jan;42(1):260-267. doi: 10.1016/j.rbmo.2020.09.020. Epub 2020 Sep 29. PMID 33288478
- [Background] Madendag IC, Madendag Y, Ozdemir AT. COVID-19 disease does not cause ovarian injury in women of reproductive age: an observational before-and-after COVID-19 study. Reprod Biomed Online. 2022 Jul;45(1):153-158. doi: 10.1016/j.rbmo.2022.03.002. Epub 2022 Mar 5. PMID 35523708
- [Background] Henarejos-Castillo I, Sebastian-Leon P, Devesa-Peiro A, Pellicer A, Diaz-Gimeno P. SARS-CoV-2 infection risk assessment in the endometrium: viral infection-related gene expression across the menstrual cycle. Fertil Steril. 2020 Aug;114(2):223-232. doi: 10.1016/j.fertnstert.2020.06.026. Epub 2020 Jun 17. PMID 32641214
- [Background] Youngster M, Avraham S, Yaakov O, Landau Rabbi M, Gat I, Yerushalmi G, Sverdlove R, Baum M, Maman E, Hourvitz A, Kedem A. IVF under COVID-19: treatment outcomes of fresh ART cycles. Hum Reprod. 2022 May 3;37(5):947-953. doi: 10.1093/humrep/deac043. PMID 35212741